CLINICAL TRIAL: NCT04400643
Title: Study Title: Prospective, Multicenter, Randomized, Controlled Study Comparing Efficacy and Safety of INTELLiVENT-ASV Versus Non-automated Ventilation in Adult ICU Subjects.
Brief Title: EASiVENT Study Comparing INTELLiVENT-ASV vs Non Automated Ventilation in Adult ICU Patients
Status: Terminated | Type: Interventional
Why Stopped: Sponsor decided to terminate the study, to terminate enrollment at this time is solely due to business reasons. No safety concerns related to the device have been identified which have in any way impacted the decision to stop the study.
Sponsor: Hamilton Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EASiVENT
Record Dates: First submitted 2020-05-14; First posted 2020-05-22 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Acute Respiratory Failure; Coma; Acute Respiratory Distress Syndrome (ARDS); Chronic Obstructive Pulmonary Disease (COPD); Obesity
MeSH Terms: conditions — Coma; Respiratory Distress Syndrome; Pulmonary Disease, Chronic Obstructive; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (2):
- INTELLiVENT-ASV (Experimental): INTELLiVENT-ASV is a software accessory that automatically adjusts ventilation and oxygenation variables to keep the patient within clinician-set target ranges, from intubation until extubation.
  Interventions: Device: INTELLiVENT-ASV
- Non-Automated ventilation (Active Comparator): In conventional ventilation modes, clinicians adjust and modify the oxygenation and ventilation parameters manually.
  Interventions: Device: Non-automated ventilation

INTERVENTIONS:
Device: INTELLiVENT-ASV — INTELLiVENT-ASV is software accessory that automatically adjust ventilation and oxygenation variables to keep the patient within clinician-set target ranges.
  Arms: INTELLiVENT-ASV
Device: Non-automated ventilation — In conventional ventilation modes, clinicians adjust and modify the oxygenation and ventilation parameters manually.
  Arms: Non-Automated ventilation

SUMMARY:
The purpose of the study is to assess the safety and efficacy of INTELLiVENT-ASV (Adaptive Support Ventilation) in adult ICU patients comparing to non automated ventilation.

DETAILED DESCRIPTION:
EASiVENT is a prospective, multicenter, randomized (1:1), Controlled Study. This study is single-blind because only the subject will be unaware of the ventilation modality administered. The reference treatment used for comparison is a combination of controlled modes for passive subjects (volume control or pressure control) and assisted/spontaneous modes for active subjects (synchronized intermittent mechanical ventilation or pressure support)

ELIGIBILITY:
Inclusion Criteria:

* Weight greater than 40 kg
* Under invasive ventilation
* Expected to be mechanically ventilated after enrollment for at least 24 hours
* Agrees to not participate in other interventional research studies involving mechanical ventilation for the duration of study
* Signature of the informed consent by the patient or his/her next-of-kin according to country or state regulation.

Exclusion Criteria:

* Fulfilling weaning criteria according to the weaning procedure of the ICU
* Need for "rescue therapy" (e.g: ECMO)
* Brain death status
* Respiratory drive disorder (Cheyne-Stokes breathing)
* Arterial hypoxia due to a non-pulmonary condition (right-to-left shunting due to congenital disease, hepato-pulmonary syndrome, )
* Broncho-pleural fistula
* Chronic or acute dyshemoglobinemia: eg.: acute CO poisoning
* Chronic respiratory failure requiring long term invasive ventilation;
* Moribund patient
* Patient under guardianship, deprived of liberties
* Any other condition, that in the opinion of the IoR/designee, would preclude informed consent (by the spouse/next of kin), make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* Low quality index on the SpO2 (Oxygen Saturation Measured by Pulse Oximetry) measurement
* Patients already enrolled in the present study in a previous episode of acute respiratory failure
* High PaCO2 - ETCO2 gap (> 2.6 kPa or 19.5 mmHg) for > 3 hours
* Patient tracheostomized at the time of inclusion
* Patient ventilated with helium

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Universitário de Lisboa Central, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Customized [Median (Inter-Quartile Range); unit: years] | 64 [25 to 75] | 67 [25 to 75] | 65 [25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 17 | 18 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Measured as Percentage of Time Spent in Optimal Range
Description: Objective of this study is to compare the efficacy of the investigational automated ventilation (INTELLiVENT-ASV) with a control ventilation group (conventional non-automated ventilation) in ICU subjects. The hypothesis is that INTELLiVENT-ASV is better than conventional non-automated ventilation in terms of efficacy. Efficacy endpoints are composite endpoints & are based on six variables that will be continuously recorded during the study period: These 6 variables: tidal volume, respiratory rate, end tidal CO2, SpO2, maximum inspiratory pressure, and maximum inspiratory pressure minus positive end-expiratory pressure. Each breath was analyzed and the breath was considered as optimal when all six variables were within predefined optimal ranges
Time Frame: up to 7 days after enrollment
Measure: Median (Inter-Quartile Range); unit: percentage of time in optimal ranges
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
percentage of time in optimal ranges | 28 [19 to 37] | 29 [8 to 39]

2. Primary Outcome: Safety Measured as Percentage of Time Spent in Sub-optimal Range
Description: Objective of this study is to compare the safety of the investigational automated ventilation (INTELLiVENT-ASV) with a control ventilation group (conventional non-automated ventilation) in ICU subjects. The hypothesis is that INTELLiVENT-ASV is better than conventional non-automated ventilation in terms of safety. Safety endpoints are composite endpoints & are based on six variables that will be continuously recorded during the study period: sub-optimal range: tidal volume, respiratory rate, end tidal CO2, SpO2, maximum inspiratory pressure, and maximum inspiratory pressure minus positive end-expiratory pressure. Each breath was analyzed and the breath was considered as sub-optimal when at least one of the six variables was within predefined sub-optimal ranges.
Time Frame: 7 days after enrollment.
Measure: Median (Inter-Quartile Range); unit: percentage of time in sub-optimal range
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
percentage of time in sub-optimal range | 16 [3 to 39] | 13 [8 to 19]

3. Secondary Outcome: Fraction of Inspiration Oxygen (FiO2) (%)
Description: FiO2 was measured breath-by-breath for all the study periods.
Time Frame: up to 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: percentage of inspired oxygen
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
percentage of inspired oxygen | 31 [27 to 38] | 36 [33 to 46]

4. Secondary Outcome: Expiratory Time Constant (s)
Description: Expiratory time constant was calculated breath-by-breath as the ratio of volume divided by flow at 75% of the expired volume.
Time Frame: up to 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: second (s)
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
second (s) | 0.59 [0.46 to 0.72] | 0.54 [0.44 to 0.65]

5. Secondary Outcome: Positive End-Expiratory Pressure (PEEP) (cm H2O)
Description: PEEP was measured breath-by-breath for all the study period.
Time Frame: up to 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: Cm H2O
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
Cm H2O | 7.7 [6.7 to 10.9] | 8.0 [5.9 to 10.3]

6. Secondary Outcome: Tidal Volume (ml)
Description: Tidal volume was measured breath-by-breath for all the study period.
Time Frame: up to 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: milliliter (ml)
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
milliliter (ml) | 420 [358 to 482] | 422 [366 to 477]

7. Secondary Outcome: Tidal Volume mL/kg Ideal Body Weight (IBW)
Description: Tidal volume mL/kg ideal body weight (IBW) will be assessed automatically breath-by-breath
Time Frame: up to 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: ml/kg of ideal body weight (IBW)
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
ml/kg of ideal body weight (IBW) | 6.8 [5.8 to 8.1] | 6.6 [5.9 to 7.1]

8. Secondary Outcome: Ventilation - Respiratory Rate
Description: Respiratory rate was measured breath-by-breath for all the study period.
Time Frame: up to 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: breath/min
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
breath/min | 20 [18 to 24] | 22 [20 to 25]

9. Secondary Outcome: Numbers of Manual Settings Changes Per Day
Description: The total number of automatic setting changes was recorded during the study period. Automatic settings included inspiratory pressure, pressure support, respiratory rate, PEEP, and inspired oxygen fraction.
Time Frame: up to 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: manual setting changes per day
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
manual setting changes per day | 12 [7 to 15] | 28 [16 to 117]

10. Secondary Outcome: Automatic Settings Changes Per Day
Description: as for outcome 9
Time Frame: up to 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: automatic setting changes per day
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
automatic setting changes per day | 1040 [511 to 1441] | 0 [0 to 0]

11. Other Pre Specified Outcome: Mortality at 28 Days (n (%))
Time Frame: up to 28 days after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
Participants | 7 | 11

12. Other Pre Specified Outcome: Duration Invasive Mechanical Ventilation (Days)
Description: Mechanical ventilation duration was recorded from the date of intubation to the date of last extubation or death if the patient died while still intubated.
Time Frame: up to 28 days from enrollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
days | 4.7 [3.0 to 8.9] | 5.3 [3.9 to 9.9]

13. Other Pre Specified Outcome: Passive Ventilation Duration (h)
Description: Passive ventilation is defined when the percentage of subject's triggered breath is lower than 25% of total respiratory rate.
Time Frame: up to 28 days from enrollment
Measure: Median (Inter-Quartile Range); unit: hours (h)
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
hours (h) | 52 [15 to 88] | 42 [6 to 92]

14. Other Pre Specified Outcome: Ventilator Free Days at Day 28 (d)
Time Frame: up to 28 days from enrollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
days | 20 [0 to 24] | 18 [0 to 22]

15. Other Pre Specified Outcome: Percentage of Time in Allocated Mode (%)
Description: The percentage of time in the allocated mode was calculated breath-by-breath according to the ventilation mode used.
Time Frame: up to 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
percentage | 100 [99 to 100] | 100 [100 to 100]

16. Other Pre Specified Outcome: Efficacy Measured as Percentage of Time Spent in Optimal Range
Description: Percentage of time spent in optimal range was calculated breath-by-breath during all the study period. Breath were classified as optimal when all six variables were in predefined optimal range: tidal volume, respiratory rate, end tidal CO2, SpO2, maximum inspiratory pressure, and maximum inspiratory pressure minus positive end-expiratory pressure.
Time Frame: up to 28 days from enrollment
Measure: Median (Inter-Quartile Range); unit: percentage of time in optimal ranges
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
percentage of time in optimal ranges | 22 [7 to 49] | 27 [8 to 59]

17. Other Pre Specified Outcome: Safety Measured as Percentage of Time Spent in Sub-optimal Range
Description: Percentage of time spent in sub-optimal range was calculated breath-by-breath during all the study period. Breath were classified as sub-optimal when at least one variable was in predefined sub-optimal range: tidal volume, respiratory rate, end tidal CO2, SpO2, maximum inspiratory pressure, and maximum inspiratory pressure minus positive end-expiratory pressure.
Time Frame: up to 28 days from enrollment
Measure: Median (Inter-Quartile Range); unit: percentage of time in sub-optimal ranges
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
Number analyzed (Participants) | 31 | 31
percentage of time in sub-optimal ranges | 30 [9 to 65] | 21 [6 to 45]

ADVERSE EVENTS:
Time Frame: up to 28 days after enrollment
Description: The study includes a general ICU patient population in need of mechanical ventilation for at least 24hrs. This population includes critically ill patients spanning a variety of primary and secondary medical conditions that can cause AEs including severe disability and death irrespective of study participation. All deaths, Serious Adverse Events, and Other Adverse Events that occurred in the study are reported in the Adverse Event module
Arm/Group | INTELLiVENT-ASV | Non-Automated Ventilation
All-Cause Mortality (participants affected / at risk) | 7/31 | 11/31
Serious Adverse Events (participants affected / at risk) | 6/31 | 5/31
Other Adverse Events (participants affected / at risk) | 2/31 | 4/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTELLiVENT-ASV (N=31) | Non-Automated Ventilation (N=31)
ACCIDENTAL EXTUBATION BY THE PATIENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 3 (3)
Cecum perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMODYNAMIC INSTABILITY IN THE CONTEXT OF DISTRIBUTIVE SHOCK (REASON FOR ADMISSION (Cardiac disorders) | 1 (1) | 0 (0)
STUDY PRINCIPAL INVESTIGATOR DECIDES TO CHANGE THE VENTILATION MODE ALLOCATED BY RANDOMIZATION (Surgical and medical procedures) | 1 (1) | 0 (0)
HYPOXIC BRAIN INJURY (Nervous system disorders) | 0 (0) | 1 (1)
HEMODYNAMIC INSTABILITY (Cardiac disorders) | 1 (1) | 0 (0)
SIGNIFICANT HYPOXEMIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUSPICION OF SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTELLiVENT-ASV (N=31) | Non-Automated Ventilation (N=31)
Ventilator-associated pneumonia (VAP) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ATELECTASIS OF LEFT LUNG (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DESOBSTRUCTION FIBROSCOPY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Barotrauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Faulty Spo2 Sensor (Product Issues) | 0 (0) | 1 (1)
MULTIPLE PERIODS OF VENT DESYNCHRONY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Premature termination resulted in a small sample size, preventing the execution of statistical analysis due to the limited number of participants in each group. The findings presented solely rely on the continuous recording of ventilator variables. Consequently, certain data captured in the electronic Case Report Form (eCRF) intended for secondary analysis, including plateau pressure, driving pressure, and blood gas results, were not taken into account.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT04400643/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT04400643/SAP_001.pdf